CLINICAL TRIAL: NCT05594108
Title: Ultrasound-guided Intrauterine Device Insertion During Family Medicine Residency
Brief Title: Ultrasound-guided IUD Insertion During Family Medicine Residency Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Angela Baerwald, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DAFM-ARB001
Record Dates: First submitted 2020-03-25; First posted 2022-10-26 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: IUD Insertion Complication
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Control group=non ultrasound guided IUD insertion Experimental group=ultrasound guided IUD insertion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Ultrasound guided IUD insertion
  Interventions: Diagnostic Test: ultrasonography
- Control Group (No Intervention): Non ultrasound guided IUD insertion

INTERVENTIONS:
Diagnostic Test: ultrasonography — transabdominal ultrasonography
  Arms: Experimental Group

SUMMARY:
The objective of this pilot study is to test that hypothesis that ultrasound guided IUD placement by family medicine residents improves patient pain scores, procedure completion time, and procedure complication rates. The secondary objective is to test the hypothesis that ultrasound guided IUD placement improves resident confidence in performing the procedure. A prospective, randomized controlled pilot study will be conducted in the Department of Academic Family Medicine at the University of Saskatchewan. All women undergoing IUD placement (hormonal or non-hormonal) at West Winds Primary Care Center from Mar 1, 2020- Mar 1, 2021 will be invited to participate. Informed consent will be obtained from each patient and the resident inserting the IUD prior to initiating study procedures. The control group will comprise 20 women undergoing non-ultrasound guided IUD placement. The experimental group will comprise 20 women undergoing transabdominal ultrasound guided IUD placement. Patient pain scores and resident confidence scores will be tabulated using likert scales and compared between control and experimental groups using independent sample t-tests. Procedure completion time (minutes) will be compared between groups using t-tests. Procedure complications rates will be categorized as: a) inability to penetrate the cervix, b) improper location, c) inability to release the IUD from the insertion device, d) perforation, e) vasovagal reactions, and f) post-procedure infection; outcomes will be compared between groups using Chi-square analyses.

ELIGIBILITY:
Inclusion Criteria:

* all women of pre or perimenopausal age undergoing IUD (hormonal or non-hormonal) placement at West Winds Primary Care Center from Mar1, 2020 to Mar1, 2021

Exclusion Criteria:

* pregnancy, < 6 weeks postpartum

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Individuals that identify as a female gender will be eligible to participate
Enrollment: 40 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
post procedure pain score | 3 years
  patient pain, likert scale

SECONDARY OUTCOMES:
procedure completion time | 3 years
  time to complete IUD insertion, mins
procedure complications | 3 years
  a) inability to penetrate the cervix, b) improper location, c) inability to release the IUD from the insertion device, d) perforation, e) vasovagal reactions, and f) post-procedure infection
residency confidence with procedure | 3 years
  family medicine resident confidence with inserting IUDs, , likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- West Winds Primary Care Center, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared, on a case by case basis, at the discretion of the principal investigator.